CLINICAL TRIAL: NCT00380107
Title: Estimation of Volume Deficit in Patients Prior to Surgery
Brief Title: Volume Deficit Prior to Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Henrik Kehlet, Section of surgical pathophysiology
Other Study IDs: Opt. medium 1
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Hypovolemia; Surgery
Keywords: Minor surgery; Volume optimization; Volume deficit; Epidural anesthesia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
It is the purpose of the researchers to identify the variation in intravascular deficits which can have relevance in high risk patients for minor and medium sized surgery.

The investigators will also estimate fluid deficit in healthy, non-fasting subjects for comparison.

DETAILED DESCRIPTION:
Intravascular volume optimization has shown to improve outcome after surgery. In minor and medium surgery , however, the preoperative volume deficit has not been estimated with functional parameters. Patient scheduled for minor surgery are included. After the patient is anesthetized the intravascular volume is optimized by stroke volume maximization by colloid boluses. Stroke volume is obtained by esophageal Doppler technique which is a minimally invasive method.

The volume estimated for optimization is considered as the functional volume deficit.

In the healthy subjects the probe will be placed in the awake subject. A standardized meal and fluid intake secures that the subjects are in a non-fasting state.

ELIGIBILITY:
Inclusion Criteria:

* Planned minor or medium sized surgery

Exclusion Criteria:

* Oesophageal pathology
* Age >90 yr or < 18 yr
* Alcohol abuse,
* Insulin dependent DM

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients for surgery in 3 procedures:
  * mastectomy
  * rad. prostatectomy
  * open adb. surgery
  And 20 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bundgaard-Nielsen, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, ABD centret, anaesthesiological dept. 2041, Copenhagen, Denmark

REFERENCES:
- [Derived] Bundgaard-Nielsen M, Jorgensen CC, Kehlet H, Secher NH. Normovolemia defined according to cardiac stroke volume in healthy supine humans. Clin Physiol Funct Imaging. 2010 Sep;30(5):318-322. doi: 10.1111/j.1475-097X.2010.00944.x. Epub 2010 Jun 10. PMID 20545713